CLINICAL TRIAL: NCT02580253
Title: Adjuvant Chemotherapy Based on the Adenosine Triphosphate Tumor Chemosensitivity
Brief Title: Adjuvant Chemotherapy Based on the Adenosine Triphosphate Tumor Chemosensitivity Assay for Hepatocellular Carcinoma After Liver Transplantation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no patients enrolled
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Weijia Fang, MD, Director, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZYYYMedOncoLT02
Record Dates: First submitted 2015-10-17; First posted 2015-10-20 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2017-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized Chemotherapy (Experimental): Two drug combination adjuvant chemotherapy based on the Adenosine Triphosphate Tumor Chemosensitivity(Oxaliplatin, Gemcitabine, Irinotecan, Paclitaxel,docetaxel, Fluorouracil,Doxorubicin,Cisplatin)
  Interventions: Drug: Individualized Chemotherapy
- mFOLFOX6 (Active Comparator): Oxaliplatin (85 mg/m2 )+Fluorouracil (2800 mg/m2 ) q2w
  Interventions: Drug: mFOLFOX6

INTERVENTIONS:
Drug: Individualized Chemotherapy — Two drug combination adjuvant chemotherapy based on the Adenosine Triphosphate Tumor Chemosensitivity(Oxaliplatin, Gemcitabine, Irinotecan, Paclitaxel,docetaxel, Fluorouracil,Doxorubicin,Cisplatin)
  Arms: Individualized Chemotherapy
Drug: mFOLFOX6 — Oxaliplatin,Fluorouracil
  Arms: mFOLFOX6

SUMMARY:
This study is a randomized, open-label, controlled study that will explore the efficacy of individualized adjuvant chemotherapy based on the adenosine triphosphate tumor chemosensitivity assay for patients with hepatocellular carcinoma after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had experienced liver transplantation with histologically confirmed advanced hepatocellular carcinoma with more one risk factor (tumour burden >8 cm, AFP>400 ng/mL,poorly differentiated,vessels invasion )
* No extrahepatic metastasis confirmed with computed tomography (CT) or magnetic resonance imaging (MRI)
* Additional inclusion criteria were age 18 years or older
* Karnofsky performance status (KPS) of at least 70%
* Adequate renal function, defined as creatinine clearance greater than 30 mL/min)
* Adequate hepatic function, defined as ALT and AST less than 5× upper limit of normal
* Adequate bone marrow function, defined as platelets greater than 100×10E9/L and WBC greater than 3.5×10E9/L.

Exclusion Criteria:

* The presence of any severe concomitant disease that could interrupt the planned treatment; intractable pain
* Hypersensitivity to study drugs
* Serious cardiovascular disease (eg, unstable coronary artery disease or myocardial infarction within 4 weeks of study start)
* National Cancer Institute CommonToxicity Criteria (NCI-CTC) grade 3 or 4 sensory or motor neuropathy
* Prior or concurrent malignancy (other than pancreatic cancer)
* Female, pregnancy or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Desease free Survival | 3 years

SECONDARY OUTCOMES:
Overall Survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- First affiliated hospital, Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Lin HS, Wan RH, Gao LH, Li JF, Shan RF, Shi J. Adjuvant chemotherapy after liver transplantation for hepatocellular carcinoma: a systematic review and a meta-analysis. Hepatobiliary Pancreat Dis Int. 2015 Jun;14(3):236-45. doi: 10.1016/s1499-3872(15)60373-3. PMID 26063023